CLINICAL TRIAL: NCT02265900
Title: Exercise and Parkinson's Disease: The Basis for Motor and Cognitive Benefits
Brief Title: Parkinson's Disease Exercise TMS PET Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Covid Restrictions have impacted longitudinal assessments for the effect of the intervention
Sponsor: Pacific Parkinson's Research Centre (Other)
Responsible Party: Principal Investigator, A. Jon Stoessl, Director of Clinical PET, Pacific Parkinson's Research Centre
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H14-02200
Record Dates: First submitted 2014-10-11; First posted 2014-10-16 (Estimated); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Parkinson Disease
Keywords: Positron Emission Tomography; Dopamine; Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise 1 (Active Comparator): One type of exercise
  Interventions: Other: Exercise
- Exercise 2 (Placebo Comparator): A different type of exercise
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — One type of exercise
  Arms: Exercise 1
Other: Exercise — A different type of exercise
  Arms: Exercise 2

SUMMARY:
The therapeutic effects of exercise in Parkinson's disease (PD) are commonly reported, however the mechanisms are unknown. The purpose of this study is to investigate the potential mechanisms of exercise in the brain for the treatment of PD.

DETAILED DESCRIPTION:
Positron Emission Tomography will be used to measure dopamine neuron density, endogenous dopamine release and neuroimflammation. We will also use functional magnetic resonance imaging (fMRI) to measure brain activity. Assessments will be conducted before and after a 12-week exercise intervention and 3-year follow-up. Participants will be randomly allocated into either an aerobic or a stretching intervention. Clinical measures of motor function, cognition and mood will also be assessed.

ELIGIBILITY:
Inclusion Criteria: Diagnosed with Parkinson's Disease, Exercise less than 3x per week.

Exclusion Criteria. Describe which potential participants will be excluded from participation, and list the criteria for their exclusion.

1. atypical Parkinson syndrome (progressive supranuclear palsy, multiple system atrophy, drug-induced etc.);
2. significant osteoporosis or arthritis;
3. other neurological disease/complications (e.g. myopathy, stroke, brain lesion, MS);
4. self-reports claustrophobia;
5. history of cancer within 5 years of study participation;
6. high dose of radiation from other procedures within the year;
7. not able to tolerate being off PD medication for up to 24 hours;
8. a female subject who is breast-feeding or pregnant.
9. Subjects who regularly use anti-inflammatories (only excluded for PBR scans).

Exclusion criteria for MRI scanning and magnetic stimulation from repetitive Transcranial Magnetic Stimulation (rTMS) scanning includes:

1. artificial heart valve;
2. brain aneurysm clip;
3. electrical stimulator for nerves or bones;
4. ear or eye implant;
5. implanted drug infusion pump;
6. coil, catheter, or filter in any blood vessel;
7. orthopedic hardware (artificial joint, plate, screws);
8. other metallic prostheses;
9. shrapnel, bullets, or other metal fragments;
10. surgery or tattoos (including tattooed eyeliner) in the last six weeks;
11. brain surgery
12. have a cardiac pacemaker, wires or defibrillator;
13. have had an injury where a piece of metal lodged in the eye or orbit;
14. have a ferromagnetic aneurysm clip; and
15. have a history of seizures/epilepsy
16. history of severe or uncontrolled headaches/migraines
17. taking medications that lower seizure threshold (e.g. amitryptiline, haloperidol)

Subjects may be excluded following study enrollment if they meet any of the following exclusion criteria:

1. significant cognitive impairment or depression;
2. significant or unstable cardiovascular or respiratory disease - all subjects will undergo a screening exercise bicycle stress test; or
3. failure to comply with the exercise or stretching intervention program by not completing at least 30 of the 36 exercise classes.
4. Severe/multiple head trauma(s)

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2014-11; Primary Completion 2020-03-12 (Actual); Study Completion 2020-03-12 (Actual)

PRIMARY OUTCOMES:
Change in Dopamine release measured by RAC PET | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: A.J. Stoessl, MD, Principal Investigator — Pacific Parkinson's Research Centre
Locations (1):
- Pacific Parkinson's Research Centre, Vancouver, British Columbia, Canada